CLINICAL TRIAL: NCT01796522
Title: Utility of Tocolytic Therapy for Maintenance Tocolysis in the Management of Threatened Preterm Delivery
Acronym: UTM/2012
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: have been published new studies that it showed the ineffectiveness of the treatments proposed in this study.
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTM/2012
Record Dates: First submitted 2013-02-14; First posted 2013-02-21 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Preterm Delivery.
MeSH Terms: conditions — Premature Birth | interventions — Progesterone; Nifedipine

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Nifedipine (60 mg / day orally) (Active Comparator): The name of this arm is Nifedipine. These Prolonged release tablets(Oros) presents a release system for 24h, acting as an osmotic pump releasing the nifedipine through an orifice in the tablet produced by laser technology.The Nifedipine tablet 60mg administered once daily to week 34 of gestation.
  Interventions: Drug: nifedipine (60 mg / day orally)
- Progesterone 200 mg / day vaginally (Active Comparator): The name of this arm is Progesterone. Soft gelatin capsule vaginal use, used in clinical practice as maintenance tocolytic therapy after episode of threatened preterm labor. The 200mg capsule administered once daily to week 34 of gestation. The patients assigned to this arm will begin treatment while the patient assigned to the arm of nifedipine.
  Interventions: Drug: progesterone 200 mg / day vaginally

INTERVENTIONS:
Drug: progesterone 200 mg / day vaginally
  Arms: Progesterone 200 mg / day vaginally
Drug: nifedipine (60 mg / day orally)
  Arms: Nifedipine (60 mg / day orally)

SUMMARY:
Hypothesis: Both nifedipine or progesterone are widely used in clinical practice as maintenance tocolytic therapy after an episode of threatened preterm delivery. Nevertheless, there is insufficient evidence to justify its routine use. The present study aims to evaluate the efficacy and safety of these tocolytic drugs for maintenance tocolysis in the management of threatened preterm delivery.

Materials and methods:

Phase III clinical trial, which evaluates the efficacy and safety of nifedipine and progesterone as maintenance tocolytic therapy until the 34th week of pregnancy in randomized women after an episode of threatened preterm delivery.

Pregnant women with singleton pregnancies are going to be evaluated, with intact membranes and cervical length less than or equal to 25 mm, which have received acute tocolysis with atosiban. They will be randomized to receive maintenance tocolysis with nifedipine (60 mg / day orally) or progesterone (200 mg / day vaginally) until week 34 of gestation. Therefore all included patients will receive treatment with proven but not agreed efficacy, to decrease the recurrence of threatened preterm delivery, prolongation of gestation and subsequent better perinatal outcome. During the course of pregnancy, patients will be monitored in outpatient obstetrics, thus checking an adequate compliance. Monitoring will continue until the end with the delivery and collection of newborn data.

The study will be single-blind, since there will be a blind evaluator. The drugs or treatments not allowed before and / or during the clinical trial are those which are indicated in the data sheet for each drug. If the patient takes antihypertensive treatment and continues it during pregnancy, dose adjustment will be done if it is needed.

Data will be collected in the case report data (CRD). The end of the test will be considered when the last recruited patient complete the gestation (delivered vaginally or cesarean), and all data from newborn are collected. If a serious adverse event occurs in a patient, the woman will immediately finish the clinical trial and will be followed until complete resolution of the episode.

Treatment is going to be considered effective if the birth occurs after 37 weeks of pregnancy with satisfactory perinatal outcome. The drugs are going to be considered safe if they do not cause adverse events in pregnant women, or if they are not serious.

Number of Subjects: 50 pregnant women

Diagnosis and main criteria for inclusion and exclusion:

Inclusion Criteria

* Pregnant women with singleton pregnancies and intact membranes which have passed an episode of threatened preterm delivery (uterine contractions with cervical change) successfully treated with atosiban as acute tocolytic therapy.
* Cervical length ≤ 25 mm. Exclusion Criteria
* ≥ 3 cm cervical dilation, multiple pregnancy, maternal medical contraindication to tocolysis with nifedipine, atosiban or progesterone, or obstetric contraindication to tocolytic treatment (severe preeclampsia, intrauterine infection, placental abruption, fetal abnormality incompatible with life, fetal death) .

Investigational product, dose and mode of administration: After a successful treatment of acute preterm labor with atosiban, is will be compared the safety and efficacy of maintenance tocolytic therapy with nifedipine 60 mg / day orally or progesterone 200 mg / day vaginally.

Therapeutic group: C08CA05 Nifedipine. G03DA04 micronized progesterone.

Route of administration: nifedipine orally. Progesterone vaginally.

Dose: Nifedipine 60 mg / day. Progesterone 200 mg / day.

Duration of treatment: From the resolution of acute episode of threatened preterm labor until 34 weeks of gestation.

Reference treatment, dose and mode of administration: Current evidence questions the utility of maintenance tocolytic therapy. No reference treatment is currently defined.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with singleton pregnancies and intact membranes which have passed an episode of threatened preterm delivery (uterine contractions with cervical change) successfully treated with atosiban as acute tocolytic therapy.
* Cervical length ≤ 25 mm.

Exclusion Criteria:

* ≥ 3 cm cervical dilation, multiple pregnancy, maternal medical contraindication to tocolysis with nifedipine, atosiban or progesterone, or obstetric contraindication to tocolytic treatment (severe preeclampsia, intrauterine infection, placental abruption, fetal abnormality incompatible with life, fetal death)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
The present study aims to evaluate the efficacy of these tocolytic drugs for maintenance tocolysis in the management of threatened preterm delivery. | 12 months

SECONDARY OUTCOMES:
The present study aims to evaluate the safety of nifedipine and progesterone as tocolytic drugs for maintenance tocolysis in the management of threatened preterm delivery. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari y Politécnic La Fe, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046